CLINICAL TRIAL: NCT00697944
Title: Ambisome® Preemptive Treatment of Multiple Colonizations by Candida in Intensive Care Patients With a Sepsis
Brief Title: Ambisome® Preemptive Treatment of Multiple Candida Colonization in Sepsis Patients
Acronym: AMBIDEX
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fovea (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: DREYFUS Medical director, FOVEA
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AMBIDEX; EUDRA-CT 2007-004444-71
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Last update posted 2008-06-16 (Estimated); Status verified 2009-03

CONDITIONS: Sepsis; Candida
Keywords: FUNGAL INFECTION; SEPSIS; INTENSIVE CARE; AMBISOME; PREEMPTIVE TREATMENT; Sepsis with candida colonisation
MeSH Terms: conditions — Sepsis; Torulopsis; Mycoses | interventions — Liposomes; liposomal amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Amphotericine in liposome (Ambisome®) — 2 IV infusions separated by one week 10 mg/kg per injection

SUMMARY:
To assess the safety of Ambisome 10 mg/kg/week in patients as a preemptive treatment in intensive care patients with a sepsis and rising candida colonisation.

Preemptive treatment (i.e., prophylactic treatment with two high doses of Ambisome® administered with an interval of one week, in patiens with a high risk of developing a fungal infection) should decrease the incidence of actual systemic infections.

The incidence of such actual fungal infections will be assessed directly and its impact on patients' survival and intensive care resourches assessed

ELIGIBILITY:
Inclusion Criteria:

* Supportive mechanical ventilation for more than 48 h
* LOD > 5 with with ailing body systems
* Candida colonisation of at least one site in addition to the digestive tract
* Suspected nosocomial infection with antibiotic treatment
* Informed consent

Exclusion Criteria:

* Patients treated with oral or systemic antifungal agents within 15 days prior to inclusion
* Patients requiring treatment with an antifungal agent or with a documented (proven or probable) fungal infection according to the EORTC criteria
* Patients with a SAPS score > 65
* Patients with neutropenia of that underwent a bone marrow tar organ transplant or with cancer chemotherapy
* Blood creatinine > 220 µmol/L
* Hemodyalysis
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-02 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Global assessment of severity of adverse events; incidence, severity and consequences of treatment emergent effects | 28-day observation period

SECONDARY OUTCOMES:
Duration of stay in the intensive care unit; occurrence of a systemic fungal infection | 28 days after first treatment administration

CONTACTS AND LOCATIONS:
Overall Officials: Elie AZOULAY, MD PhD, Principal Investigator — University Teaching Hospital Saint Louis, Paris
Locations (2):
- France (2):
  - Chu Michallon, Grenoble
  - Hopital Saint Louis, Paris

REFERENCES:
- [Derived] Azoulay E, Timsit JF, Lautrette A, Legriel S, Max A, Ruckly S, Misset B, Cohen Y, Wolff M. Weekly high-dose liposomal amphotericin B (L-AmB) in critically ill septic patients with multiple Candida colonization: The AmBiDex study. PLoS One. 2017 May 22;12(5):e0177093. doi: 10.1371/journal.pone.0177093. eCollection 2017. PMID 28531175